CLINICAL TRIAL: NCT00237172
Title: Phase II Clinical Study of Imatinib Mesylate in Patients With Malignant Gastrointestinal Stromal Tumors (Extension Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571B1202
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; Imatinib; STI571; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (1):
- Imatinib Mesylate (Experimental): 400 mg once daily
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — once daily
  Other Names: STI571

SUMMARY:
This is a extension study of CSTI571B1201 study

ELIGIBILITY:
Inclusion Criteria:

- Patients who completed the CSTI571B1201 study

Exclusion Criteria:

-

Other protocol-defined inclusion / exclusion criteria may apply.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2002-09; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
To study the antineoplastic effect of the investigational drug.

SECONDARY OUTCOMES:
To study the safety and pharmacokinetics of the investigational drug.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals